CLINICAL TRIAL: NCT03889678
Title: Utility of Color-flow Doppler to Identify Peripheral Intravenous Catheter Infiltration in Adult Surgical Patients
Brief Title: Color Doppler and Peripheral Venous Catheters
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor, Augusta University
Other Study IDs: 1237593
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Extravasation; Vein Injury
Keywords: Color flow Doppler; infiltration; extravasation; peripheral intravenous catheters; general anesthesia
MeSH Terms: interventions — Echocardiography, Doppler, Color

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral IV: Patients with peripheral intravenous line in place undergoing elective surgery
  Interventions: Diagnostic Test: Color flow doppler

INTERVENTIONS:
Diagnostic Test: Color flow doppler — Color flow doppler proximal to vein insertion site to document flow

SUMMARY:
Objective: To evaluate color Doppler flow ultrasound compared to standard clinical techniques, to detect the correct position of peripheral intravenous catheters in adult surgical patients.

Methods: A prospective study is conducted in adult (>18 years old) patients scheduled to undergo elective surgery. Peripheral intravenous catheter position is evaluated with standard clinical techniques (free flow of fluid from a hanging bag, easy saline injection, and aspiration of blood), and with color flow Doppler ultrasound proximal to the insertion site. Comparative test performance is carried out.

DETAILED DESCRIPTION:
Confirmation of adequate peripheral intravenous catheter placement should be determined before using the parenteral route; however, there is no gold standard universally accepted for this purpose. Determination of the correct position of freshly inserted peripheral intravenous catheters and already established intravenous lines depends largely on subjective clinical signs such as visual evidence of swelling around the insertion site, low resistance to infusion and free back-flow of blood. Ultrasound-guided cannulation of peripheral veins has gained popularity in recent years and is standard of practice in some institutions. Primarily used in guiding central line placement, the applications of ultrasound for vascular access continue to expand in the perioperative setting, thanks to its easy use, non-invasiveness and safety profile. On the other hand, utilization of color Doppler technology with flow injection test has been shown to be a valuable tool for early recognition of malfunctioning intravenous catheters. The color Doppler flow technique is both safe and reliable, and aids in identification of correct intravascular position of venous catheters in children.

This study aims to test the hypothesis that the color Doppler flow technique is superior to standard clinical techniques (free flow from a hanging intravenous fluid bag, aspiration of venous blood with syringe, and non-obstructed hand injection of 2 mL of normal saline) to detect the correct position of peripheral intravenous catheters in adult surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years undergoing elective surgery with an indwelling peripheral venous catheter.

Exclusion Criteria:

* Patients with open wounds in the vicinity of the intravenous line insertion site or scar tissue on the extremity, as well as those with dressings, bandages, or casts on the extremity precluding adequate use of ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with a peripheral venous catheter in situ, scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Intravascular catheter position | 2 minutes
  Confirmation of adequate position of peripheral vein catheter confirmed by color flow Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided